CLINICAL TRIAL: NCT03895905
Title: Comparison of Cervical Pathologies in the Presence of High Risk Hpv Positivity in Normal Women With Cytology
Brief Title: Comparison of Cervical Pathologies in the Presence of High Risk Hpv Positivity
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.7.03
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Human Papilloma Virus; Cervical Neoplasm
Keywords: colposcopy; High Risk HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Genotype of HR-HPV 16/18: Patients with genotype of HR-HPV 16/18 who underwent cervical biopsy with colposcopy
  Interventions: Diagnostic Test: colposcopy and colposcopic biopsy
- Genotype of HR-HPV Non-16/18: Patients with genotype of HR-HPV non-16/18 who underwent cervical biopsy with colposcopy
  Interventions: Diagnostic Test: colposcopy and colposcopic biopsy

INTERVENTIONS:
Diagnostic Test: colposcopy and colposcopic biopsy — high-risk hpv positivity and colposcopy and cervical biopsy results will be evaluated. thus, it will be defined whether colposcopy will be performed routinely at high-risk hpv.

SUMMARY:
The only malignancy screening test among gynecological cancers is cervical cancer.

Cytology examination and Hpv typing with smear are used as screening tests. Hpv positivity is detected in more than 90% of cervical cancers. However, only the Hpv 16-18 type positive patients undergo colposcopy in the routine screening program.

Patients with Smear negative, Type 16-18 high-risk Hpv positivity are evaluated by quota after 1 year.

the authors performed colposcopy with this study; authors aimed to compare the results of patients with type 16-18 Hpv positivity and type 16-18 high-risk Hpv positivity and to find out whether there was any difference between them.

In this way, other high-risk Hpv types other than type 16-18 (31,33,35,45,51, etc.) may be exposed to premalign cervical lesions and possible cancer in a number of earlier and earlier periods by performing colposcopic examination instead of expecting to perform quota after 1 year. we aimed to remove.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years old
* patients with normal smear

Exclusion Criteria:

* Patients with invasive cervical cancer,
* HIV-positive patients,
* ASCUS and more risky premalignant lesions in cytology,
* Over the age of 65 and
* Patients under 20 years of age,
* patients with another known gynecological malignancy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk HPV and colposcopy were the study groups.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Genotype of HR-HPV 16/18 | 1 MONTH
  Results of colposcopies and retrieved colposcopic biopsy of patients with Genotype of HR-HPV 16/18
Genotype of HR-HPV non 16/18 | 1 MONTH
  Results of colposcopies and retrieved colposcopic biopsy of patients with Genotype of HR-HPV non 16/18

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)